CLINICAL TRIAL: NCT00889863
Title: A Randomized, Double-blind, Placebo Controlled, Withdrawal Study of Flare Prevention of Canakinumab (ACZ885) in Patients With Systemic Juvenile Idiopathic Arthritis (SJIA) and Active Systemic Manifestations
Brief Title: Flare Prevention Study of Canakinumab in Patients With Active Systemic Juvenile Idiopathic Arthritis (SJIA)
Acronym: β-SPECIFIC 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Pediatric Rheumatology International Trials Organization (Other)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CACZ885G2301; EudraCT: 2008-005479-82
Record Dates: First submitted 2009-04-21; First posted 2009-04-29 (Estimated); Results first posted 2012-10-16 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-09

CONDITIONS: Systemic Juvenile Idiopathic Arthritis With Active Flare
Keywords: Flare; arthritis; IL-1beta antagonist; systemic juvenile idiopathic arthritis; Juvenile rheumatoid
MeSH Terms: conditions — Arthritis; Arthritis, Juvenile | interventions — canakinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Canakinumab (Experimental): In Part I participants received open label 4 mg/kg canakinumab subcutaneous injection every 4 weeks for up to 32 weeks. For the first 8 weeks Part Ia (4 weeks) and Ib (4 weeks) patients maintained a stable oral steroid dose (prednisone or equivalent) followed by Ic an up to 20 week steroid tapering period and then Id a 4 week stable steroid dose period. Participants were then randomized to receive either 4 mg/kg canakinumab subcutaneous injection or placebo comparator in Part II and remained on the stable oral steroid dose for 24 weeks. At 24 weeks in Part II participants with a >0.2 mg/kg and ≤ 0.5 mg/kg and no flare could restart steroid tapering. If the steroid dose was ≤ 0.2 mg/kg participants continued to maintain their current dose for the remainder of Part II.
  Interventions: Drug: canakinumab
- Placebo (Placebo Comparator): Participants in Part II received placebo matching canakinumab subcutaneous injection every 4 weeks. At 24 weeks in Part II participants with a >0.2 mg/kg and ≤0.5 mg/kg and no flare could restart steroid tapering. If the steroid dose was ≤0.2 mg/kg participants continued to maintain their current dose for the remainder of Part II.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: canakinumab — Canakinumab 4 mg/kg dose subcutaneous injection supplied as 6 mL glass vials each containing 150 mg canakinumab as a lyophilized cake.
  Arms: Canakinumab
Drug: placebo — Placebo powder matching canakinumab supplied as 6 mL glass vials containing a lyophilized cake for subcutaneous injection every 4 weeks in Part II.
  Arms: Placebo

SUMMARY:
This two-part study assessed the sustained efficacy of canakinumab in the double-blind Part II and the ability to taper steroids in the open label Part I.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of systemic juvenile idiopathic arthritis as per International League Against Rheumatism (ILAR) definition that must have occurred at least 2 months prior to enrollment with onset of disease < 16 years of age.

  -Arthritis in one or more joints with or preceded by fever of at least 2 weeks duration that is documented to be daily for at least 3 days with accompanying symptoms
* Active disease at the time of enrollment defined as follows:

  * At least 2 joints with active arthritis (using American College of rheumatology) ACR definition of active joint)
  * Documented spiking, intermittent fever (body temperature > 38oC) for at least 1 day during the screening period within 1 week before first study drug dose
  * C-reactive protein > 30 mg/L (normal range < 10 mg/L)
* No concomitant use of second line agents such as disease-modifying and/ or immunosuppressive drugs will be allowed with the exception of:

  * Stable dose of methotrexate for at least 8 weeks prior to the screening visit, and/or folic/folinic acid per standard medical practice
  * Stable dose of no more than one non-steroidal anti-inflammatory drug for at least 2 weeks prior to the screening visit
  * Stable dose of steroid treatment < or = to 1.0 mg/kg/day in 1-2 doses per day of oral prednisone or equivalent

Exclusion criteria:

* Diagnosis of active macrophage-activation syndrome (MAS) within the last 6 months
* Risk factors for tuberculosis
* Patients with active or recurrent bacterial, fungal or viral infection at the time of enrollment, including patients with evidence of HIV infection, Hepatitis B and Hepatitis C infection

Other protocol inclusion/exclusion criteria may apply

Ages: 2 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 177 (Actual)
Dates: Start 2009-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (73):
- United States (12):
  - Arkansas Children's Hospital Research Inst, Little Rock, Arkansas
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Louisville, Louisville, Kentucky
  - New England Medical Center - Department of Allergy, Boston, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts
  - St Barnabas Ambulatory Care Center, Livingston, New Jersey
  - Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital/Neurology, Cincinnati, Ohio
  - Legacy Emanuel Hospital, Portland, Oregon
  - Legacy Emanual Research, Portland, Oregon
  - Specially For Children, Austin, Texas
- Argentina (3):
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Capital Federal
  - Novartis Investigative Site, La Plata
- Belgium (4):
  - Novartis Investigative site, Brussels
  - Novartis Investigative site, Ghent
  - Novartis Investigative Site, Laken
  - Novartis Investigative site, Leuven
- Brazil (4):
  - Novartis Investigative Site, Curitiba
  - Novartis Investigative site, Porto Alegre
  - Novartis Investigative site, Rio de Janiero
  - Novartis Investigative site, São Paulo
- Canada (4):
  - Novartis Investigative site, Vancouver, British Columbia
  - Novartis Investigative site, Halifax, Nova Scotia
  - Novartis Investigative site, Toronto, Ontario
  - Novartis Investigative site, Montreal, Quebec
- France (4):
  - Novartis Investigative Site, Le Kremlin-Bicêtre
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Strasbourg
- Germany (9):
  - Novartis Investigative Site, Bad Bamstedt
  - Novartis Investigative site, Berlin
  - Novartis Investigative Site, Bremen
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Geißen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Saint Augustin
  - Novartis Investigative Site, Stuttgart
- Novartis Investigative Site, Budapest, Hungary
- Israel (5):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Kfar Saba
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Rehovot
- Italy (9):
  - Novartis Investigative Site, Bologna
  - Novartis Investigative Site, Florence
  - Novartis Investigative Site, Genova
  - Novartis Investigative site, Milan
  - Novartis Investigative site, Napoli
  - Novartis Investigative site, Padua
  - Novartis Investigative site, Rome
  - Novartis Investigative site, Scafati
  - Novartis Investigative site, Torino
- Novartis Investigative site, Utrecht, Netherlands
- Novartis Investigative Site, Oslo, Norway
- Novartis Investigative Site, Lima, Peru
- Novartis Investigative site, Warsaw, Poland
- South Africa (4):
  - Novartis Investigative site, Berea, Durban
  - Novartis Investigative site, Mayville, Durban
  - Novartis Investigative site, Johannesburg
  - Novartis Investigative site, Pretoria
- Spain (3):
  - Novartis Investigative site, Barcelona
  - Novartis Investigative site, Madrid
  - Novartis Investigative site, Valencia
- Novartis Investigative site, Stockholm, Sweden
- Switzerland (3):
  - Novartis Investigative Site, Bern
  - Novartis Investigative site, Lausanne
  - Novartis Investigative site, Zurich
- Turkey (Türkiye) (3):
  - Novartis Investigative site, Ankara
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir

REFERENCES:
- [Derived] Ruperto N, Brunner HI, Quartier P, Constantin T, Wulffraat NM, Horneff G, Kasapcopur O, Schneider R, Anton J, Barash J, Berner R, Corona F, Cuttica R, Fouillet-Desjonqueres M, Fischbach M, Foster HE, Foell D, Radominski SC, Ramanan AV, Trauzeddel R, Unsal E, Levy J, Vritzali E, Martini A, Lovell DJ; Paediatric Rheumatology International Trials Organisation (PRINTO) and the Pediatric Rheumatology Collaborative Study Group (PRCSG). Canakinumab in patients with systemic juvenile idiopathic arthritis and active systemic features: results from the 5-year long-term extension of the phase III pivotal trials. Ann Rheum Dis. 2018 Dec;77(12):1710-1719. doi: 10.1136/annrheumdis-2018-213150. Epub 2018 Sep 29. PMID 30269054
- [Derived] Brachat AH, Grom AA, Wulffraat N, Brunner HI, Quartier P, Brik R, McCann L, Ozdogan H, Rutkowska-Sak L, Schneider R, Gerloni V, Harel L, Terreri M, Houghton K, Joos R, Kingsbury D, Lopez-Benitez JM, Bek S, Schumacher M, Valentin MA, Gram H, Abrams K, Martini A, Lovell DJ, Nirmala NR, Ruperto N; Pediatric Rheumatology International Trials Organization (PRINTO) and the Pediatric Rheumatology Collaborative Study Group (PRCSG). Early changes in gene expression and inflammatory proteins in systemic juvenile idiopathic arthritis patients on canakinumab therapy. Arthritis Res Ther. 2017 Jan 23;19(1):13. doi: 10.1186/s13075-016-1212-x. PMID 28115015
- [Derived] Grom AA, Ilowite NT, Pascual V, Brunner HI, Martini A, Lovell D, Ruperto N; Paediatric Rheumatology International Trials Organisation and the Pediatric Rheumatology Collaborative Study Group; Leon K, Lheritier K, Abrams K. Rate and Clinical Presentation of Macrophage Activation Syndrome in Patients With Systemic Juvenile Idiopathic Arthritis Treated With Canakinumab. Arthritis Rheumatol. 2016 Jan;68(1):218-28. doi: 10.1002/art.39407. PMID 26314396
- [Derived] Ruperto N, Brunner HI, Quartier P, Constantin T, Wulffraat N, Horneff G, Brik R, McCann L, Kasapcopur O, Rutkowska-Sak L, Schneider R, Berkun Y, Calvo I, Erguven M, Goffin L, Hofer M, Kallinich T, Oliveira SK, Uziel Y, Viola S, Nistala K, Wouters C, Cimaz R, Ferrandiz MA, Flato B, Gamir ML, Kone-Paut I, Grom A, Magnusson B, Ozen S, Sztajnbok F, Lheritier K, Abrams K, Kim D, Martini A, Lovell DJ; PRINTO; PRCSG. Two randomized trials of canakinumab in systemic juvenile idiopathic arthritis. N Engl J Med. 2012 Dec 20;367(25):2396-406. doi: 10.1056/NEJMoa1205099. PMID 23252526
- See also: Related Info — http://www.novartisclinicaltrials.com
- See also: Related Info — http://www.juvenilearthritisresearch.com

RESULTS

PARTICIPANT FLOW:
Period: Part I: Open Label
Arm/Group | Canakinumab | Placebo
Started | 177 | 0 (No participants received placebo in Part I.)
Entered Part Ia | 145 | 0
Entered Part Ib | 142 | 0
Entered Part Ic | 92 (Patients steroid free at study entry entered Part Id directly and did not participate in Part Ic.) | 0
Entered Part 1d | 103 | 0
Completed | 100 | 0
Not Completed | 77 | 0
Not completed — Death | 1 | 0
Not completed — Adverse Event | 4 | 0
Not completed — Unsatisfactory therapeutic effect | 72 | 0
Period: Part II: Randomized Double Blind
Arm/Group | Canakinumab | Placebo
Started | 50 | 50
Completed | 39 | 24
Not Completed | 11 | 26
Not completed — Adverse Event | 0 | 4
Not completed — Unsatisfactory therapeutic effect | 11 | 20
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Protocol deviation | 0 | 1

BASELINE CHARACTERISTICS:
Arm/Group | Canakinumab
Number analyzed (Participants) | 177
Age Continuous [Mean (Standard Deviation); unit: years] | 8.7 (4.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98
  Male | 79

OUTCOME MEASURES:

1. Primary Outcome: Part I: Percentage of Patients Who Were on Steroids at Entry Into Part I and Who Were Able to Taper Steroid as Per Protocol in at Least 25% of the Patients Who Entered the Study Taking a Steroid
Description: Ability to taper oral steroids: if dose reduced from start of Part I to end of Part Ic from > 0.8 mg/kg/day to ≤ 0.5 mg/kg/day, or from ≥ 0.5 mg/kg/day and ≤ 0.8 mg/kg/day by at least 0.3 mg/kg, or from any initial dose to ≤ 0.2 mg/kg/day, while maintaining a minimum adapted ACR 30 pediatric criterion. Patients on oral steroids at study entry who did not enter Part 1c are considered steroid tapering failures.
Time Frame: 32 Weeks
Population: Participants from the Full Analysis Set who were taking oral steroids at the beginning of Part I.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 128
Percentage of participants | 44.5 [37.1 to 52.2]

2. Primary Outcome: Part II: Survival Estimate of Time to Flare
Description: Kaplan Meier estimate of the probability to experience a flare. Flare was defined as at least 1 of the following.
  * Reappearance of fever (>38°C, lasting for at least 2 consecutive days) not due to infections
  * Flare according to the JIA pediatric criteria for flare (all criteria must have been met):
  * ≥ 30% worsening in at least 3 of the first 6 response variables
  * ≥ 30% improvement in not more than 1 of the first 6 response variables Patients who discontinued the study while in Part II were counted as flared unless they discontinued because of inactive disease for at least 24 weeks in Part II.
Time Frame: Part II was event driven. The study was stopped when the required number of 37 flares had occurred (88 weeks)
Population: Full Analysis Set in Part II
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 50 | 50
Days | NA [NA to NA] — Not observed. Less than 50% participants with a flare. | 236.0 [141.0 to 449.0]

3. Secondary Outcome: Part I: Percentage of Patients on Steroids at Study Start Who Reached a Steroid Dose ≤0.2 mg/kg at End of Part Ic
Time Frame: 28 Weeks
Population: Participants from the Full Analysis set who were taking oral steroids at the start of the study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 128
Percentage of participants
  steroid free | 32.8 [24.8 to 41.7]
  >0 and ≤ 0.2 mg/kg/day | 18.8 [12.4 to 26.6]

4. Secondary Outcome: Part I: Percentage of Participants on Steroids at the Start of 1c Who Were Able to Taper Steroids by the End of Part 1c
Time Frame: Start of Part Ic (After Week 8) to End of Part Ic (Week 28)
Population: Participants from the Full Analysis set who were taking oral steroids at the start of Part Ic.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 92
Percentage of participants | 62.0 [52.9 to 70.4]

5. Secondary Outcome: Part I: Percentage of Participants With Minimum American College of Rheumatology (ACR) 30/50/70/90/100 at the End of Part I
Description: Adapted ACR Pediatric 30/50/70/90/100 criteria are defined as meeting all of the following:
  * improvement from baseline of ≥ 30%, ≥ 50%, ≥ 70%, ≥ 90%, or 100%, in at least 3 of the first 6 response variables
    1. Physician's global assessment of disease activity
    2. CHAQ-patient's overall well-being
    3. CHAQ-Functional ability
    4. # of joints with active arthritis
    5. # of joints with limitation of motion
    6. C-Reactive Protein.
  * no intermittent fever in the preceding week
  * no more than one of the first 6 response variables worsening by more than 30%
Time Frame: Baseline, 32 Weeks
Population: Participants from the full analysis set with an assessment at the given time-point.
Measure: Number; unit: Percentage of participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 175
Percentage of participants
  Non-Responders | 22.9
  ACR 30 Response | 77.1
  ACR 50 Response | 73.1
  ACR 70 Response | 64.6
  ACR 90 Response | 51.4
  ACR 100 Response | 34.3

6. Secondary Outcome: Part I: Time to First Minimum American College of Rheumatology (ACR50) and Normal C-Reactive Protein
Description: Duration in days in the study to the first minimum adapted ACR Pediatric 50 criteria and a normal (<10mg/L) C-Reactive Protein
Time Frame: Baseline, Week 32
Population: Participants from the Full Analysis Set Part I with ACR 50 and a Normal CRP.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Canakinumab
Number analyzed (Participants) | 63
Days | 20.4 (8.7)

7. Secondary Outcome: Part I: Time to First Minimum American College of Rheumatology (ACR70) and Normal C-Reactive Protein
Description: Duration in days in the study to the first minimum adapted ACR Pediatric 70 criteria and a normal (<10mg/L) C-Reactive Protein
Time Frame: Baseline, Week 32
Population: Participants from the Full Analysis Set Part I with ACR 70 and a Normal CRP.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Canakinumab
Number analyzed (Participants) | 65
Days | 24.5 (21.58)

8. Secondary Outcome: Part I: Percentage of Participants With Body Temperature ≤ 38 Degrees Celsius at Day 3 in Part 1a
Time Frame: Day 3
Population: Participants from the Full Analysis Set Part I with temperature readings at Day 3.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 141
Percentage of participants | 98.6 [95.0 to 99.8]

9. Secondary Outcome: Part II: Survival Analysis of Time to a Worsening in American College of Rheumatology (ACR) Response
Description: Kaplan Meier estimate of the time in days to the probability of worsening of the ACR response.
  ACR response is determined by the following items:
  1. Physician's global assessment of disease activity
  2. CHAQ-patient's overall wellbeing
  3. CHAQ-Functional ability
  4. Number of joints with active arthritis
  5. Number of joints with limitation of motion
  6. C-Reactive Protein.
  7. No intermittent fever in the preceding week
Time Frame: Part II was event driven. The study was stopped when the required number of 37 flares had occurred (88 weeks)
Population: Full Analysis Set Part II
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 50 | 50
Days | NA [171.0 to NA] — Not observed as less than 50% of patients had a worsening of ACR response. | 141.0 [85.0 to 281.0]

10. Secondary Outcome: Part I: Change in Disability Over Time in the Child Health Assessment Questionnaire-Disability Index (CHAQ-DI) From Baseline to End of Part I
Description: The childhood health assessment questionnaire, CHAQ was used to assess physical ability and functional status of patients as well as quality of life. The disability dimension consists of 20 multiple choice items concerning difficulty in performing eight common activities of daily living; dressing and grooming, arising, eating, walking, reaching, personal hygiene, gripping and other "activities". Parents choose from four response categories, ranging from 0(without any difficulty) to 3(unable to do). A negative change indicates improvement.
Time Frame: Baseline, End of Part I (Week 32)
Population: Participants from the Full Analysis Set Part I with data at baseline and End of Part I.
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | Canakinumab
Number analyzed (Participants) | 175
Score on a scale | -0.8750 (0.86492) [-2.875 to 1.125]

11. Secondary Outcome: Part II: Change in Disability Over Time by the Child Health Assessment Questionnaire-Disability Index (CHAQ-DI)
Description: CHAQ-DI assessed physical ability and functional status of patients and quality of life. 20 multiple choice items concerning difficulty in performing 8 common activities of daily living; dressing and grooming, arising, eating, walking, reaching, personal hygiene, gripping and other "activities". Parents choose from 4 response categories, ranging from 0(without any difficulty) to 3(unable to do).
  Repeated measures Analysis of Covariance with treatment group, visit day, prednisone (or equivalent) dose and adapted ACR 70 response reached at the end of Part Id as covariates.
Time Frame: Start of Part II (Week 32), End of Part II ( total duration-88 weeks)
Population: Full Analysis set Part II.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 50 | 50
Score on a scale | 0.1184 (0.17592) | 0.1258 (0.18241)

12. Secondary Outcome: Part I: Change in Health Related Quality of Life Over Time by Child Health Questionnaire (CHQ-PF50)
Description: The CHQ-PF50© is an instrument used to measure Health Related Quality of Life in children 5-18 from the parent's perspective. The questionnaire measures the following concepts: Physical functioning, Role/social emotional, Role/social behavior, Role/social physical, Bodily pain, General behavior, Mental health, Self-esteem, General health perception, Change in health, Parental impact - emotional, Parental impact - time, Family activities, and Family cohesion. Summaries are provided for Physical Health and Psychosocial Health. Scores range from 0-100. Increase in score represents improvement.
Time Frame: Baseline, End of Part I ( Week 32)
Population: Participants from the Full Analysis Set Part I-age 5 to 18 years.
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | Canakinumab
Number analyzed (Participants) | 125
Score on a scale
  Physical Health Score | 21.8050 (16.10377) [-21.554 to 62.309]
  Psychosocial Health Score | 8.2223 (11.50688) [-21.710 to 38.854]

13. Secondary Outcome: Part II: Change in Health Related Quality of Life Over Time by Child Health Questionnaire (CHQ-PF50)
Description: CHQ-PF50 measures Physical functioning, Role/social emotional, behavior and physical, Bodily pain, General behavior, Mental health, Self-esteem, General health perception, Change in health, Parental impact-emotional, Parental impact-time, Family activities and cohesion. Summaries are provided for Physical Health and Psychosocial Health. An increase in score indicates improvement. Repeated measures Analysis of Covariance change from start of Part II with treatment group, visit day, prednisone(or equivalent) dose and adapted ACR70 Pediatric response reached at the end of Part Id as covariates.
Time Frame: Start Part II (Week 32), End Part II (total duration - 88 Weeks)
Population: Full Analysis Set Part II-patients aged 5-18 years.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 39 | 37
Score on a scale
  Physical Health Score | 3.9 (2.54) | -0.3 (2.53)
  Psychosocial Health Score | 2.5 (1.88) | -0.5 (1.86)

ADVERSE EVENTS:
Groups:
- Canakinumab: Part I: In Part I participants received open label 4 mg/kg canakinumab subcutaneous injection every 4 weeks for up to 32 weeks. For the first 8 weeks Part Ia (4 weeks) and Ib (4 weeks) patients maintained a stable oral steroid dose (prednisone or equivalent) followed by Ic an up to 20 week steroid tapering period and then Id a 4 week stable steroid dose period.
- Canakinumab: Part II: Participants received 4 mg/kg canakinumab subcutaneous injection in Part II and remained on the stable oral steroid dose for 24 weeks. At 24 weeks in Part II participants with a >0.2 mg/kg and ≤ 0.5 mg/kg and no flare could restart steroid tapering. If the steroid dose was ≤ 0.2 mg/kg participants continued to maintain their current dose for the remainder of Part II.
- Placebo: Part II: Participants in Part II received placebo matching canakinumab subcutaneous injection every 4 weeks. At 24 weeks in Part II participants with a >0.2 mg/kg and ≤0.5 mg/kg and no flare could restart steroid tapering. If the steroid dose was ≤0.2 mg/kg participants continued to maintain their current dose for the remainder of Part II.
Arm/Group | Canakinumab: Part I | Canakinumab: Part II | Placebo: Part II
Serious Adverse Events (participants affected / at risk) | 15/177 | 6/50 | 6/50
Other Adverse Events (participants affected / at risk) | 138/177 | 40/50 | 35/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab: Part I (N=177) | Canakinumab: Part II (N=50) | Placebo: Part II (N=50)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 3 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
Medical device complication (General disorders) | 1 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 1 | 0 | 0
Adenovirus infection (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0
Gastrointestinal viral infection (Infections and infestations) | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0
Lymph node abscess (Infections and infestations) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1
C-reactive protein increased (Investigations) | 1 | 0 | 0
Coagulation test abnormal (Investigations) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 1 | 0
Platelet count increased (Investigations) | 1 | 0 | 0
Serum ferritin increased (Investigations) | 1 | 0 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0
Juvenile arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Histiocytosis haematophagic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Measles (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Haptoglobin decreased (Investigations) | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Splenic neoplasm malignancy unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 1
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab: Part I (N=177) | Canakinumab: Part II (N=50) | Placebo: Part II (N=50)
Nasopharyngitis (Infections and infestations) | 27 | 7 | 7
Headache (Nervous system disorders) | 23 | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 20 | 8 | 6
Pyrexia (General disorders) | 18 | 7 | 5
Upper respiratory tract infection (Infections and infestations) | 18 | 6 | 5
Vomiting (Gastrointestinal disorders) | 18 | 1 | 4
Abdominal pain (Gastrointestinal disorders) | 17 | 6 | 4
Diarrhoea (Gastrointestinal disorders) | 17 | 1 | 3
Rhinitis (Infections and infestations) | 17 | 5 | 7
Gastroenteritis (Infections and infestations) | 14 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 12 | 5
Abdominal pain upper (Gastrointestinal disorders) | 9 | 2 | 2
Eczema (Skin and subcutaneous tissue disorders) | 9 | 3 | 1
Nausea (Gastrointestinal disorders) | 9 | 3 | 1
Pharyngitis (Infections and infestations) | 9 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 6 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0
Oral herpes (Infections and infestations) | 3 | 4 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 4 | 2
Tinea pedis (Infections and infestations) | 0 | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 3
Seasonal allergy (Immune system disorders) | 0 | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.